CLINICAL TRIAL: NCT00498342
Title: The Effect of Administration on N-Acetylcysteine on Serum Creatinine Levels in Patients With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: FlowMedic (Industry)
Responsible Party: Dr. Richard Solomon, University of Vermont
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: UVM07-205
Record Dates: First submitted 2007-07-06; First posted 2007-07-10 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2007-07

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: N-acetylcysteine

SUMMARY:
Primary outcome: Serum creatinine change at 4 hours and 48 hours following 4 doses of N-acetylcysteine (total 4800 mg) compared to baseline serum creatinine.

Secondary outcome: Serum Cystatin C change at 4 hours and 48 hours post 4 doses of N-acetylcysteine compared to baseline serum Cystatin C.

DETAILED DESCRIPTION:
N-acetylcysteine has been reported to lower serum creatinine in normal individuals. The mechanism of this effect is unknown but possible stimulation of tubular secretion of creatinine has been hypothesized based upon a lack of effect on Cystatin C levels. If this effect also occurs in subjects with chronic kidney disease, interpretation of clinical trials using N-acetylcysteine for prophylaxis of acute kidney injury would be confounded. To answer whether such confounding occurs, 50 patients with stable chronic kidney disease (Stage 3-5) will be given 4 doses of N-acetylcysteine, 1200 mg each, with measurement of serum creatinine and Cystatin C before, 4 hours and 48 hours after the last dose. No other interventions, including changes in medications, will be permitted during the study.

ELIGIBILITY:
Inclusion Criteria:

* Estimated GFR 10-59 ml/min/1.73m2 by 4 variable MDRD equation
* Less than a 10% difference between the baseline creatinine and the recruitment creatinine obtained within 3 months of the trial

Exclusion Criteria:

* Unable to give informed consent
* Unwillingness to return for follow-up blood sampling
* Unstable renal function
* Subjects taking H2-blockers

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-06; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Serum creatinine change at 4 hours and 48 hours following 4 doses of N-acetylcysteine (total 4800 mg) compared to baseline serum creatinine | 48 hours

SECONDARY OUTCOMES:
Serum Cystatin C change at 4 hours and 48 hours post 4 doses of N-acetylcysteine compared to baseline serum Cystatin C | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Solomon, M.D., Principal Investigator — University of Vermont/Fletcher Allen Health Care,Inc.
Locations (1):
- University of Vermont /Fletcher Allen Health Care, Inc., Burlington, Vermont, United States

REFERENCES:
- [Background] Solomon R. Contrast media nephropathy--how to diagnose and how to prevent? Nephrol Dial Transplant. 2007 Jul;22(7):1812-5. doi: 10.1093/ndt/gfm207. Epub 2007 Apr 20. No abstract available. PMID 17449491
- [Background] Solomon RJ, Natarajan MK, Doucet S, Sharma SK, Staniloae CS, Katholi RE, Gelormini JL, Labinaz M, Moreyra AE; Investigators of the CARE Study. Cardiac Angiography in Renally Impaired Patients (CARE) study: a randomized double-blind trial of contrast-induced nephropathy in patients with chronic kidney disease. Circulation. 2007 Jun 26;115(25):3189-96. doi: 10.1161/CIRCULATIONAHA.106.671644. Epub 2007 Jun 11. PMID 17562951
- [Background] Solomon R, Deray G; Consensus Panel for CIN. How to prevent contrast-induced nephropathy and manage risk patients: practical recommendations. Kidney Int Suppl. 2006 Apr;(100):S51-3. doi: 10.1038/sj.ki.5000375. No abstract available. PMID 16612402
- [Background] Solomon R, Barrett B. Follow-up of patients with contrast-induced nephropathy. Kidney Int Suppl. 2006 Apr;(100):S46-50. doi: 10.1038/sj.ki.5000374. PMID 16612401
- [Background] Solomon R, Briguori C, Bettmann M. Selection of contrast media. Kidney Int Suppl. 2006 Apr;(100):S39-45. doi: 10.1038/sj.ki.5000373. PMID 16612400